CLINICAL TRIAL: NCT03320174
Title: Single Site, Randomized, Double Blind, Placebo-Controlled Study to Assess the Long-Term Safety of Tafenoquine
Brief Title: Long-Term Safety Study of Tafenoquine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: 60 Degrees Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 60PH04
Record Dates: First submitted 2017-10-18; First posted 2017-10-25 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2020-01

CONDITIONS: Healthy Volunteers
Keywords: tafenoquine; australia
MeSH Terms: interventions — tafenoquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Identically matched placebo control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tafenoquine 200 mg (2 x 100 mg tablets) (Active Comparator): Tafenoquine 200 mg (2 x 100 mg tablets) daily for three consecutive days, followed by study treatment (tafenoquine 200 mg or placebo) once per week for 51 weeks
  Interventions: Drug: Tafenoquine
- Placebo (Placebo Comparator): Placebo daily for three consecutive days, followed by study treatment (tafenoquine 200 mg or placebo) once per week for 51 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tafenoquine — Tafenoquine 200mg
  Arms: Tafenoquine 200 mg (2 x 100 mg tablets)
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This randomized, double-blind, placebo controlled study will involve 600 healthy (Glucose-6-Phosphate Dehydrogenase [G6PD] normal) volunteers. Participants who meet the eligibility criteria will be randomized (ratio 1:1) to receive a loading dose of either tafenoquine 200 mg (2 x 100 mg tablets) or placebo daily for three consecutive days, followed by study treatment (tafenoquine 200 mg or placebo) once per week for 51 weeks, with safety follow-up visits at Weeks 4, 12, 24, and 52. All participants will return to the clinic at Week 64 for an end of study visit. If the participant has an ongoing AE at the Week 64 visit will continue to be assessed for up to 3 more times at approximately 12-week intervals or until resolution or stabilization of the AE whichever is earlier.

ELIGIBILITY:
Main Inclusion Criteria:

1. Completion of the written informed consent process (signed).
2. Male or female age 18 to 55 years inclusive, in good health as assessed by the Investigator.
3. Normal G6PD enzyme activity levels as defined by the parameters of the specific G6PD test employed at the local laboratory.
4. Negative HBsAg and HCV, HIV-1, HIV-2 antibody screen at the screening visit.
5. Negative serum pregnancy test.
6. Use acceptable method of birth control.
7. Hematology, biochemistry and urinalysis results at screening that are within the local laboratory reference range or, if outside the range, not clinically significant as judged by the Investigator in accordance with approved clinically acceptable laboratory ranges, documented prior to study start.
8. Willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Main Exclusion Criteria:

1. History of allergy or intolerance to tafenoquine, primaquine or any excipients.
2. History of thalassemia or current or past history of methemoglobinemia or methemoglobin >2% at screening.
3. History of eye disease or surgery
4. Having previously received hydroxychloroquine for skin conditions or rheumatological diseases, chloroquine for malaria, tamoxifen, amiodarone or other drugs that may affect the optic nerve/retina/cornea within 30 days or 5 half-lives (whichever is longer) of study start. There are no travel restrictions, but the choice of concurrent anti-malarial must be atovaquone-proguanil if the participant chooses to take a registered antimalarial drug while travelling.
5. Any current diagnosis of Axis I psychiatric disorders

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Proportion of Subjects with Spectral Domain Optical Coherence Tomography (SD-OCT) and Quantitative Fundus Auto Fluorescence (qFAF) with clinically significant changes compared with baseline. | After 12 months of exposure to study drug

SECONDARY OUTCOMES:
The incidence, severity and relationship to the investigational medicinal product of AEs | After 12 months of exposure to study drug
Mean change from baseline in key SD OCT parameters including central subfield thickness, total macular volume, and parafoveal (inner ring of Early Treatment Diabetic Retinopathy Study, and retinal thickness | After 12 months of exposure to study drug
Proportion of participants with ellipsoid or interdigitating zone disruption | After 12 months of exposure to study drug
Mean change from baseline in Best Corrected Visual Acuity | After 12 months of exposure to study drug
Proportion of participants with corneal deposits from slit lamp examination of the corneal epithelium | After 12 months of exposure to study drug
Proportion of participants with new abnormalities compared with baseline observed with color retinal digital photography | After 12 months of exposure to study drug
Proportion of participants with new abnormalities compared with baseline observed with multifocal electroretinography | After 12 months of exposure to study drug
Proportion of participants with new abnormalities compared with baseline observed with microperimetry | After 12 months of exposure to study drug
Proportion of participants with any clinically significant change in ETDRS BCVA (defined as >15 letter change [≥ 3 lines] of change in ETDRS BCVA at 4 meters) | After 12 months of exposure to study drug
Proportion of participants who develop a color deficiency using the Farnsworth-Munsell 100 (FM-100) hue test | After 12 months of exposure to study drug
Proportion of participants who develop a loss of 0.12 or greater logarithm of contrast sensitivity (logCS) on the Mars letter contrast sensitivity test | After 12 months of exposure to study drug
Proportion of participants with any new anomaly on the backlit ETDRS chart | After 12 months of exposure to study drug
Proportion of participants who develop a psychiatric disorder in accordance with DSM-5 as assessed with the Mini International Neuropsychiatric Interview (M.I.N.I.) 7.0.2 assessment questionnaire | After 12 months of exposure to study drug
Proportion of participants with an AE of dizziness or vertigo and severity as assessed by the Dizziness Handicap Inventory | After 12 months of exposure to study drug
Mean change from baseline visual analog scale score (1-100) in Getting to Sleep (GTS) as assessed by the Leeds Sleep Evaluation Questionnaire (LSEQ). | After 12 months of exposure to study drug
Mean change from baseline visual analog scale score (1-100) Quality of Sleep (QOS) as assessed by the Leeds Sleep Evaluation Questionnaire (LSEQ). | After 12 months of exposure to study drug
Mean change from baseline visual analog scale score (1-100) Awake Following Sleep (AFS) as assessed by the Leeds Sleep Evaluation Questionnaire (LSEQ). | After 12 months of exposure to study drug
Mean change from baseline visual analog scale score (1-100) Behavior Following Wakening (BFW) as assessed by the Leeds Sleep Evaluation Questionnaire (LSEQ). | After 12 months of exposure to study drug

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Retina Consultants of Southern Colorado, Colorado Springs, Colorado
  - Valley Retina Institute, McAllen, Texas
- Linear Clinical Research, Nedlands, Western Australia, Australia

REFERENCES:
- [Derived] Novitt-Moreno A, Martidis A, Gonzalez V, Ransom J, Scott CB, Dow G, Reid M, Smith B, Zottig VE, Read LT, Garver Baldwin LS, Chen FK. Long-term safety of the tafenoquine antimalarial chemoprophylaxis regimen: A 12-month, randomized, double-blind, placebo-controlled trial. Travel Med Infect Dis. 2022 Jan-Feb;45:102211. doi: 10.1016/j.tmaid.2021.102211. Epub 2021 Nov 18. PMID 34801714